CLINICAL TRIAL: NCT03632499
Title: From Research to Clinical Practice. Applying an Algorithm for Prognosis of Upper Limb Paresis in Patients With Subacute Stroke
Brief Title: An Algorithm for Prognosis of Upper Limb Paresis in Patients With Subacute Stroke
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 63518
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2018-03

CONDITIONS: Stroke; Upper Limb Hypertonia; Physical Activity
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: rehabilitation — rehabilitation

SUMMARY:
Aim study 1:Assess the accuracy of PREP2 when applied in a subacute rehabilitation setting.

Aim study 2: Prediction of real life UL use. Method: A prospective cohort study. Main outcome measure study 1: Action Research Arm Test (ARAT), measuring UL motor function.

Main outcome study 2: use ratio between affected and unaffected UL measured by accellerometer.

Secondary outcome measure: Fugl-Meyer Motor Assessment for UL (FM).

DETAILED DESCRIPTION:
Background Accurate prediction of recovery of UL function after stroke can lead to targeted rehabilitation. The Predict Recovery Potential (PREP2) algorithm combines individual prediction of UL function with recommendations for treatment. The PREP2 algorithm is based on clinical assessment of UL paresis combined with transcranial magnetic stimulation (TMS) to examine corticospinal tract integrity. For this PhD project the PREP2 is modified to be applicable in a rehabilitation setting and the initial assessment of PREP2, the SAFE score, is carried out at day 14.

Study 1 Aim: Assess the accuracy of PREP2 when applied in a subacute rehabilitation setting.

Hypothesis: PREP2 applied at day 14 post stroke accurately predicts UL function 3 months after stroke for a minimum of 75 % of the patients.

Method: A prospective cohort study. Setting and population: The study will take place at Hammel Neurorehabilitation Centre and University Research Clinic. Ninety patients will be included.

Inclusion criteria: First or recurrent ischemic or hemorrhagic stroke (diagnosis verified by CT or MR scan); New upper limp impairment; Less than 15 days post stroke; ≥ 18 years; Able to follow simple commands and cooperate with examinations Main outcome measure: Action Research Arm Test (ARAT), measuring UL motor function.

Secondary outcome measure: Fugl-Meyer Motor and sensory Assessment for UL. Functional Independence Measure (FIM).

Examined at baseline: Pain wil be assessed with a verbal rating scale. Inferior subluxation in the glenohumoral joint. Neglect will be assessed with star cancellation test and line bisection test

Study 2 Prediction of real life UL use Hypothesis: PREP2 can be used to predict real life UL use 3 months post stroke. Patients: The entire cohort from study 1 will be included. Real life use will be assessed with accelerometers at 3 months follow up.

Main outcome: is the use ratio between affected and unaffected UL.

ELIGIBILITY:
Inclusion Criteria:

* First or recurrent ischemic or hemorrhagic stroke (diagnosis verified by CT or MR scan)
* New upper limp impairment; Less than 15 days post stroke
* ≥ 18 years
* Able to follow simple commands and cooperate with examinations

Exclusion Criteria:

* Subarachnoid hemorrhages
* UL motor residuals from former stroke
* Severe illness with life expectancy < 6 months
* Place of residence more than 1½ hours drive away and not reachable for follow up assessments
* Patients with contraindications for TMS are excluded from the TMS part of the study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stroke in a rehabilitation setting
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Action Research Arm test | dec 2019
  Upper limb function test

SECONDARY OUTCOMES:
Fugl Meyer Motor and sensory assesment | Dec 2019
  Upper limb function test
Accellerometry | dec 2019
  accellerometer

CONTACTS AND LOCATIONS:
Overall Officials: Iris Brunner, phd, Study Chair — Iris.Brunner@rm.dk
Locations (1):
- Camilla Lundquist, Hammel, Denmark

IPD SHARING:
Plan to Share IPD: No